CLINICAL TRIAL: NCT01079247
Title: A Randomized Clinical Trial of Restrictive vs. Traditional Blood Transfusion Practices in Burn Patients
Brief Title: A Trial of Restrictive Versus Traditional Blood Transfusion Practices in Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Burn Association (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABA-MCTG-0001
Record Dates: First submitted 2010-02-26; First posted 2010-03-03 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Burn Injury
Keywords: Burn; Transfusion; blood; hemoglobin
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal (Active Comparator): Maintain hemoglobin at 10-11 g/dL
  Interventions: Other: Liberal transfusion threshold
- Restrictive (Active Comparator): Maintain hemoglobin at 7-8 g/dL
  Interventions: Other: Restrictive transfusion threshold

INTERVENTIONS:
Other: Restrictive transfusion threshold — maintain hemoglobin at 7-8 g/dL
  Arms: Restrictive
Other: Liberal transfusion threshold — Maintain hemoglobin at 10-11 g/dL
  Arms: Liberal

SUMMARY:
The purpose of this study is to find out if burn injured patients do better receiving fewer blood transfusions than what is traditionally given. We traditionally provide blood transfusions to maintain a hemoglobin level, which is an indicator of the level of red blood cells that carry oxygen in your body, to above 10 g/dl (g/dl stands for grams per deciliter and is the standard measurement used to indicate the level of red blood cells in your blood). However, a preliminary study indicated that maintaining the hemoglobin level to above 7-8 g/dl with less blood transfusion, as compared to a hemoglobin level of 10 g/dl and above, would reduce the occurrence of blood infection, duration on the respirator and length of hospital stay, yet would achieve similar survival in both groups.

ELIGIBILITY:
Inclusion Criteria:

* >20% TBSA burn with anticipated operation need on admission as determined by attending physician
* age >18 years
* Admission within 96 hours of injury

Exclusion Criteria:

* <18 years of age
* pregnancy
* inability or unwillingness to receive blood products
* history of chronic anemia (hemoglobin <9.0 g/dL one month prior to enrollment)
* preexisting need for hemodialysis
* brain death or imminent brain death
* non-survivable burn as determined by the attending burn surgeon
* angina or acute myocardial infarction
* preexisting hematologic disease
* Length of hospital stay anticipated to be < 2 weeks
* Transfusion administered at outside hospital before admit

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2010-02-28 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Blood Stream Infection | 1 week after randomization and weekly thereafter through discarge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Tina L Palmieri, MD, Principal Investigator — University of California, Davis
Locations (18):
- United States (15):
  - Maricopa Integrated Health System (Arizona Burn Center), Phoenix, Arizona
  - Arrowhead Regional Medical Center, Colton, California
  - Community Regional Medical Center, Fresno, California
  - University of California Davis Medical Center-Regional Burn Center, Sacramento, California
  - University of California, San Diego, San Diego, California
  - Washington Hospital Burn Center, Washington D.C., District of Columbia
  - University of Florida Health Science, Gainesville, Florida
  - Doctors Hospital-Joseph M Still Burn Center, Augusta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of North Carolina at Chapel Hill (Jaycee Burn Center), Chapel Hill, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Oregon Burn Center Legacy Health System, Portland, Oregon
  - University of Texas SouthWestern Medical Center, Dallas, Texas
  - U.S. Army Institute of Surgical Research (USAISR), Fort Sam Houston, Texas
  - University of Utah Intermountain School of Medicine, Salt Lake City, Utah
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Sunnybrook Health Science Center, Toronto, Ontario
- New Zealand National Burn Centre-Middlemore Hospital, Auckland, New Zealand

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Gibran NS, Shipper E, Phuong J, Braverman M, Bixby P, Price MA, Bulger EM; NTRAP Burns & Reconstructive Surgery Panel Group. Developing a national trauma research action plan: Results from the Burn Research Gap Delphi Survey. J Trauma Acute Care Surg. 2022 Jan 1;92(1):201-212. doi: 10.1097/TA.0000000000003409. PMID 34554139
- [Derived] Cartotto R, Taylor SL, Holmes JH 4th, Peck M, Cochran A, King BT, Bhavsar D, Tredget EE, Mozingo D, Greenhalgh D, Pollock BH, Palmieri TL. The Effects of Storage Age of Blood in Massively Transfused Burn Patients: A Secondary Analysis of the Randomized Transfusion Requirement in Burn Care Evaluation Study. Crit Care Med. 2018 Dec;46(12):e1097-e1104. doi: 10.1097/CCM.0000000000003383. PMID 30234568
- [Derived] Palmieri TL, Holmes JH 4th, Arnoldo B, Peck M, Potenza B, Cochran A, King BT, Dominic W, Cartotto R, Bhavsar D, Kemalyan N, Tredget E, Stapelberg F, Mozingo D, Friedman B, Greenhalgh DG, Taylor SL, Pollock BH. Transfusion Requirement in Burn Care Evaluation (TRIBE): A Multicenter Randomized Prospective Trial of Blood Transfusion in Major Burn Injury. Ann Surg. 2017 Oct;266(4):595-602. doi: 10.1097/SLA.0000000000002408. PMID 28697050